CLINICAL TRIAL: NCT07131566
Title: Immune Response in Cervical Lymph Nodes of Patients With Head and Neck Cancer
Status: Recruiting | Type: Observational
Sponsor: Lars Olaf Cardell (Other)
Responsible Party: Sponsor-Investigator, Lars Olaf Cardell, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: Vetenskapsrådet 2024-03236; K 2022-2823 (Other: Karolinska Sjukhuset)
Record Dates: First submitted 2025-06-25; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma Head and Neck Cancer (HNSCC)
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sentinel Node detection and Biopsy — Fine Needle aspiration from sentinel Lymph Nodes

SUMMARY:
Objective:

The aim of this study is to characterize the inflammatory response in patients with head and neck cancer. More specifically, the study intend to investigate inflammatory and genetic differences between the primary tumor, the sentinel lymph node, and other regional lymph nodes. The investigator also aim to assess how the immunological and genetic responses differ in lymph nodes with and without metastases.

To enable the detection of metastases in lymph nodes containing very few cancer cells, the investigator are developing a method to identify tumor cells using flow cytometry. Additionally, both tumor tissue and lymph nodes will undergo in vitro testing of checkpoint blockade therapy, a relatively new form of cancer immunotherapy.

Methods:

Biopsies from the primary tumor will be used to assess local inflammation. Fine-needle aspirates and dissected lymph node tissue will be analyzed to study inflammatory and genetic responses, as well as to detect tumor cells within these nodes. Blood samples from patients with head and neck cancer will be analyzed for inflammatory mediators.

Lymph nodes from patients without cancer will be collected during benign neck surgeries. Immunological and genetic parameters from these control lymph nodes will be compared to those from the cancer patients to identify disease-specific patterns.

DETAILED DESCRIPTION:
Statistical analyse Plan: All data will be log-transformed to approximate normal distribution. For pairwise comparisons Student's t-test will be used. For multiple comparisons one-way ANOVA followed by a suitable post-hoc test will be performed.

Power: Power has been determined based on available previous data. The investigator will have access to samples from up to 300 study subjects that can be used generate different datasets. The calculated sample size ranges from 20 to 60 samples per group depending on the specific research question. This calculation was conducted assuming two-tailed comparisons, with, significance p<0.05, and power 80%.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of primary HNSCC,
2. tumor excision combined with a sentinel node-assisted elective neck dissection or sentinel node biopsy alone performed at Karolinska University Hospital, Stockholm, Sweden
3. willingness to participate in the study.

Exclusion Criteria:

1. systematic autoimmune diseases
2. synchronous or previous second malignancies or hemo-lymphopoietic malignancies
3. any other acute or chronic condition that could influence the immunological environment in the lymph nodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HNSCC with surgery at Karolinska University Hospital, Stockholm Sweden
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of cervical lymph nodes with tumor cells detected by flow cytometry | Baseline (at surgery or biopsy)
  Flow cytometric detection of tumor cells in sentinel node, other cervical lymph nodes, or fine-needle aspirates. Reported as the percentage of examined lymph nodes containing tumor cells. Unit of measure: % of lymph nodes
Immunological cell profile in sentinel node measured by flow cytometry | Baseline (at surgery or biopsy)
  Quantification of immune cell populations (e.g., CD4+, CD8+ T cells, B cells) in sentinel node, expressed as number of cells per mg of tissue. Unit of measure: % of total cells

SECONDARY OUTCOMES:
Differential gene expression between sentinel node and non tumour draining lymph node. | Baseline (at surgery or biopsy)
  RNA sequencing of biopsies from sentinel node and non tumour draining lymph node to identify differentially expressed genes (log2 fold change, p-value).unit of measure: Fold change in gene expression

OTHER OUTCOMES:
Topographical localization of sentinel node | Baseline (pre-surgery imaging)
  SPECT-CT imaging to determine sentinel node location, reported as frequency (%) of nodes located in predefined anatomical regions. Unit of measure: % of sentinel nodes in each location

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No